CLINICAL TRIAL: NCT03878082
Title: Perioperative Regular Usage of Propacetamol to Reduce Post Cesarean Section Uterine Contraction Pain and Opioid Consumption
Brief Title: Propacetamol to Reduce Post Cesarean Section Uterine Contraction Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, attending physician, department of anesthesiology, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19MMHIS044e
Record Dates: First submitted 2019-03-07; First posted 2019-03-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Uterine Pain
Keywords: cesarean section; uterine contraction pain; propacetamol
MeSH Terms: interventions — propacetamol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propacetamol 1g (Active Comparator): pain control with IVPCA and propacetamol 1g every 6 hours for 2 days
  Interventions: Drug: Propacetamol 1g; Drug: IVPCA
- propacetamol 2g (Active Comparator): pain control with IVPCA and propacetamol 2g every 6 hours for 2 days
  Interventions: Drug: Propacetamol 2g; Drug: IVPCA
- IVPCA (Placebo Comparator): pain control with IVPCA
  Interventions: Drug: IVPCA

INTERVENTIONS:
Drug: Propacetamol 1g — pain control with IVPCA and propacetamol 1g every 6 hours for 2 days
  Other Names: Propacetamol 1g + IVPCA
  Arms: propacetamol 1g
Drug: Propacetamol 2g — pain control with IVPCA and propacetamol 2g every 6 hours for 2 days
  Other Names: Propacetamol 2g + IVPCA
  Arms: propacetamol 2g
Drug: IVPCA — pain control with IVPCA
  Other Names: IVPCA alone

SUMMARY:
To evaluate that perioperative regular usage of propacetamol to reduce post cesarean section uterine contraction pain and opioid consumption

DETAILED DESCRIPTION:
The most common method of pain control after cesarean section is intravenous patient-control analgesia (IVPCA) with morphine. Multimodal analgesia could improve the quality of perioperative pain control and reduceside effects of opioids. Previous researches marked that perioperative pain after cesarean section includes somatic wound pain and visceral uterine contraction pain.

According to Academy of Breastfeeding Medicine, propacetamol is a safe pain-killer for an expectant mother and almost free from breast milk after intravenous injection. This study is a prospective double-blind randomized-controlled trial to evaluate that propacetamol could reduce visceral uterine contraction pain after cesarean section. Post cesarean section women will divide into three groups:

1. pain control with IVPCA for 2 days
2. pain control with IVPCA and propacetamol 1g every 6 hours for 2 days
3. pain control with IVPCA and propacetamol 2g every 6 hours for 2 days

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy more than 36 weeks which is expected to receive Caesarean section
* Post Caesarean section woman, age greater than or equal to 20 years old
* ASA physical status class 1 or 2

Exclusion Criteria:

* ASA physical status class 3 or above
* Less than 20 years old
* Past caesarean section for longitudinal wounds
* Undergone major abdominal surgery
* Chronic pain
* Allergic to morphine or Propacetamol
* Liver dysfunction
* Treatment with anticoagulant
* Emergency operation

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post Caesarean section woman
Enrollment: 100 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of pain assessed by NRS | Every 8 hours from post-anesthesia care unit to 2 days after the cesarean section
  Change of pain assessed by Numerical Rating Scale: respondent selects a whole number (0-10 integers) that best reflects the intensity of the pain
Incidence of treatment-relate adverse events | Two days after the cesarean section
  the complications or side effects during intervention, such as nausea/vomiting, skin itching, GI discomfort, urinary retention, and respiratory depression
Opioid consumption | Two days after the cesarean section
  Comparison with the placebo group, the requirement of opoid

SECONDARY OUTCOMES:
Satisfaction assessed by the NRS | Two days after the cesarean section
  Participants' satisfaction about post-operative pain management assessed by Numerical Rating Scale: respondent selects a whole number (0-10 integers , dissatisfied -> satisfied) that best reflects the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valentine AR, Carvalho B, Lazo TA, Riley ET. Scheduled acetaminophen with as-needed opioids compared to as-needed acetaminophen plus opioids for post-cesarean pain management. Int J Obstet Anesth. 2015 Aug;24(3):210-6. doi: 10.1016/j.ijoa.2015.03.006. Epub 2015 Mar 23. PMID 25936786
- [Background] Ortiz MI, Ponce-Monter HA, Mora-Rodriguez JA, Barragan-Ramirez G, Barron-Guerrero BS. Synergistic relaxing effect of the paracetamol and pyrilamine combination in isolated human myometrium. Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):22-6. doi: 10.1016/j.ejogrb.2011.02.011. Epub 2011 Mar 24. PMID 21439705
- [Background] Gadsden J, Hart S, Santos AC. Post-cesarean delivery analgesia. Anesth Analg. 2005 Nov;101(5 Suppl):S62-S69. doi: 10.1213/01.ANE.0000177100.08599.C8. PMID 16334493